CLINICAL TRIAL: NCT02655185
Title: Study to Evaluate Association of Blood Lipid Levels With Atrial Fibrillation Incidence in Patients With Chronic Heart Failure
Brief Title: Novel Risk Factors of Atrial Fibrillation in Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yangzhou No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Chen, associate chief physician, Yangzhou No.1 People's Hospital
Other Study IDs: 2016003
Record Dates: First submitted 2016-01-10; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: Lipids; Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Heart failure

SUMMARY:
The purpose of this study is to determine whether lipid levels are related with incidence of atrial fibrillation in Patients with chronic heart failure.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in clinical practice. Chronic Heart failure (CHF) has become a major clinical and public health problem. Both AF and CHF often co-exist and complicate each other's administration.Several risk factors have been demonstrated to be associated with the risk of AF in Patients with CHF.

Lopez et al. found that higher levels of low-density lipoprotein cholesterol (LDLc) and total cholesterol were associated with a lower incidence of AF independently of other risk factors from the Atherosclerosis Risk in Communities (ARIC) study.

Thus the purpose of this study is to determine whether lipid levels are related with incidence of atrial fibrillation in Patients with chronic heart failure. This study maybe provide a novel opinion on the prevention of AF in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic heart failure

Exclusion Criteria:

* Use of statins

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital patients with a diagnosis of chronic heart failure will be recruited at Yangzhou No.1 people's hospital, China.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with newly emerging atrial fibrillation as assessed by electrocardiogram | three years

SECONDARY OUTCOMES:
Cardiovascular mortality | three years
Worsing heart failure assessed by decreased NYHA class and left ventricular ejection fraction | three years
rate of rehospitalization | three years

CONTACTS AND LOCATIONS:
Overall Officials: Chen - Liu, MD, Principal Investigator — Yangzhou No.1 People's Hospital

IPD SHARING:
Plan to Share IPD: No